CLINICAL TRIAL: NCT05573724
Title: A Non-randomized, Open-label, Fixed-sequence Phase I Study to Assess the Effect of Itraconazole (a CYP3A4 Inhibitor) on the Pharmacokinetics of AZD5305 in Patients With Advanced Solid Malignancies
Brief Title: Drug-drug Interaction Study With AZD5305 and Itraconazole in Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D9720C00005; 2022-001450-33 (EudraCT Number)
Record Dates: First submitted 2022-10-07; First posted 2022-10-10 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Malignancies
Keywords: Tumors; Pharmacokinetics; Itraconazole; AZD5305; Safety; Tolerability
MeSH Terms: conditions — Neoplasms | interventions — AZD5305; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Part A:
  The participants will receive a single oral dose of AZD5305 on Day 1, followed by a 2-day washout. Then Itraconazole will be dosed for 3 days [BD] on Day 4 and [OD] on Days 5 and 6, then a single oral dose of AZD5305 administered concurrently with Itraconazole on Day 7 and only Itraconazole on Days 8 to 12.
  Part B:
  Patients proceeding to Part B after completing Part A of the study will receive AZD5305 OD as monotherapy.
  Interventions: Drug: AZD5305; Drug: Itraconazole

INTERVENTIONS:
Drug: AZD5305 — In Part A, the participants will receive a single dose of AZD5305 on Day 1 and Day 7.
  In Part B, the participants will receive AZD5305 once daily.
Drug: Itraconazole — In Part A, the participants will receive Itraconazole twice daily on Day 4 and once daily on Days 5-12

SUMMARY:
This study is a single-arm, open-label, multi-centre drug-drug interaction (DDI) study of AZD5305 administered orally in patients with advanced solid tumours.

DETAILED DESCRIPTION:
This study will comprise of two study parts, Part A and Part B. Part A of the study will assess the effect of multiple doses of Itraconazole on the single dose pharmacokinetic (PK) parameters of AZD5305 which will last up to 13 days. The patients will then continue into Part B and receive AZD5305 monotherapy at the discretion of the Investigator if the patients are deemed to still derive benefit from continued treatment until disease progression.

The Part A of this study follows a non-randomized, open-label, 2-intervention design. Patients will receive the following two study interventions, AZD5305 and Itraconazole: a single oral dose of AZD5305 alone, multiple oral doses of itraconazole alone, and then a single oral dose of AZD5305 administered concomitantly with multiple doses of itraconazole.

In Part B, the patients may continue the study with AZD5305 monotherapy after completing Part A of the study. AZD5305 monotherapy will continue until disease progression, unacceptable toxicities, initiation of alternative anticancer therapy, withdrawal of consent, or other reasons to discontinue study treatment occur.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
* Males and females aged ≥ 18 years at the time of screening.
* Patients with documented evidence of locally advanced unresectable or metastatic solid tumours, excluding lymphoma, who have exhausted standard of care options (or for which no standard therapies exist) and may be suitable for AZD5305 monotherapy treatment.
* Adequate organ and marrow function.
* An Eastern Cooperative Oncology Group Performance Status (ECOG PS): 0 to 2 with no deterioration over the previous 2 weeks.
* Life expectancy ≥ 12 weeks.
* Female patients of childbearing potential. Must have a negative pregnancy test result at screening and prior to each Part of study intervention.
* Female patients must not breastfeed and must not donate or retrieve ova for their own use from screening to approximately 6 months after the last dose of study intervention.

Exclusion Criteria:

* Previous enrolment in the present study (ie, dosing with AZD5305 previously initiated in this study).
* Positive for detection of drugs of abuse or alcohol at screening.
* Concomitant use of medications or herbal supplements known to be cytochrome P450 3A4 enzyme (CYP3A4) substrates, strong, and moderate inhibitors or inducers.
* Patients with germline Breast cancer gene-mutated relapsed advanced ovarian cancer who have received three or more previous lines of chemotherapy.
* Using of proton pump inhibitors, histamine H2 receptor antagonists and other antiacid agents.
* Using of calcium channel blockers.
* Concomitant use of drugs that are known to prolong or shorten QT and have a known risk of Torsade's de Pointes (TdP).
* During the 4 weeks prior to the first dose, receiving continuous corticosteroids.
* Major surgery within 4 weeks of the first dose of study intervention.
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study intervention.
* Treatment with any of the following: any investigational agents or study interventions from a previous clinical study within 5 half-lives or 3 weeks (whichever is shorter) of the first dose of study intervention; any other anticancer treatment within the following time periods prior to the first dose of study intervention: Cytotoxic and non-cytotoxic treatment: 3 weeks or five half-lives (whichever is shorter); Biological products including immuno-oncology agents: 4 weeks before enrolment.; any live virus or bacterial vaccine within 28 days of the first dose of study intervention.
* Any concurrent anticancer therapy or concurrent use of prohibited medications.
* With the exception of alopecia, and peripheral neuropathy; any unresolved toxicities from prior therapy greater than CTCAE Grade 1.
* Any known history of persisting (> 2 weeks) severe pancytopenia.
* Spinal cord compression, or brain metastases unless asymptomatic and treated and stable and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent.
* Any evidence of severe or uncontrolled systemic diseases, including, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus.
* Patients with any known predisposition to bleeding.
* Any of the following cardiac criteria: mean resting QTcF > 450 ms or QTcF < 340 ms obtained from triplicate ECGs and averaged, recorded within 5 minutes; any factors that increase the risk of QT prolongation, shortening or risk of arrhythmic events such as hypokalaemia, congenital long or short QT syndrome, family history of long QT syndrome, familial short QT syndrome, or unexplained sudden death under 40 years of age; any clinically important abnormalities in rhythm, conduction or morphology of resting ECG eg, complete left bundle branch block, second- or third-degree atrioventricular block, and clinically significant sinus node dysfunction not treated with pacemaker.
* Other cardiovascular diseases.
* Patients with history of MDS/AML or with features suggestive of MDS/AML.
* Refractory nausea and vomiting, chronic GI diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD5305.
* Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s).
* Any condition that, in the opinion of the Investigator, would interfere with evaluation of the study intervention or interpretation of patient safety or study results.
* Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
* Uncontrolled intercurrent illness within the last 12 months.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
Part A: Area under the concentration-time curve from time zero to infinity (AUCinf) | Day 1-4, Day 7-13
  The effect of Itraconazole on the AUCinf of AZD5305 will be assessed. The ratios of geometric means of test intervention (AZD5305 + Itraconazole; parent and metabolite[s], if applicable) relative to reference intervention (AZD5305 alone) of AUCinf will be presented.
Part A: AUC from time zero to time of last measurable concentration (AUClast) | Day 1-4, Day 7-13
  The effect of Itraconazole on the AUClast of AZD5305 will be assessed. The ratios of geometric means of test intervention (AZD5305 + Itraconazole; parent and metabolite[s], if applicable) relative to reference intervention (AZD5305 alone) of AUClast will be presented.
Part A: Maximum plasma drug concentration (Cmax) | Day 1-4, Day 7-13
  The effect of Itraconazole on the Cmax of AZD5305 will be assessed. The ratios of geometric means of test intervention (AZD5305 + Itraconazole; parent and metabolite[s], if applicable) relative to reference intervention (AZD5305 alone) of Cmax will be presented.
Part A: Apparent total body clearance of drug from plasma (CL/F) | Day 1-4, Day 7-13
  The effect of Itraconazole on the PK of AZD5305 will be assessed.
Part A: Terminal elimination half-life (t½λz) | Day 1-4, Day 7-13
  The effect of Itraconazole on the PK of AZD5305 will be assessed.
Part A: Time to maximum observed concentration (Tmax) | Day 1-4, Day 7-13
  The effect of Itraconazole on the PK of AZD5305 will be assessed.
Part A: Apparent volume of distribution based on the terminal phase (Vz/F) | Day 1-4, Day 7-13
  The effect of Itraconazole on the PK of AZD5305 will be assessed.

SECONDARY OUTCOMES:
Part A and Part B: Number of participants with Adverse Events (AEs) and Serious Adverse events (SAEs) | Part A: From screening until post-treatment follow-up (28 days after last dose) (approximately 13 days if continuing into Part B); Part B: From Cycle 1 day 1 until Post treatment follow up (28 days after last dose) (approximately 12 months)
  Participants with potentially clinically significant AEs and SAEs will be determined.
Part A and Part B: Number of Participants with Laboratory Value Abnormalities and/or AEs | Part A: From screening until post-treatment follow-up (28 days after last dose) (approximately 13 days if continuing into Part B); Part B: From Cycle 1 Day 1 until Post treatment follow-up (28 days after last dose) (approximately 12 months)
  Participants with potentially clinically significant laboratory values will be determined.
Part A and Part B: Number of Participants with Vital Sign Abnormalities and/or AEs | Part A: From screening until post-treatment follow-up (28 days after last dose) (approximately 13 days if continuing into Part B); Part B: From Cycle 1 Day 1 until Post treatment follow-up (28 days after last dose) (approximately 12 months)
  Participants with potentially clinically significant vital signs values will be determined.
Part A and Part B: Number of Participants with Electrocardiogram (ECG) Abnormalities and/or AEs | Part A: From screening until post-treatment follow-up (28 days after last dose) (approximately 13 days if continuing into Part B); Part B: From Cycle 1 Day 1 until Post treatment follow-up (28 days after last dose) (approximately 12 months)
  Participants with potentially clinically significant ECG values will be determined.
Part A and Part B: Number of Participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) Abnormalities and/or AEs | Part A: From screening until post-treatment follow-up (28 days after last dose) (approximately 13 days if continuing into Part B); Part B: From Cycle 1 Day 1 until Post treatment follow-up (28 days after last dose) (approximately 12 months)
  Participants with potentially clinically significant ECOG PS values will be determined.

CONTACTS AND LOCATIONS:
Locations (2):
- Research Site, Chisinau, Moldova
- Research Site, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in a sponsor approved tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home